CLINICAL TRIAL: NCT05471505
Title: Safety and Effectiveness of Apixaban Compared to Warfarin in NVAF Patients at Higher Risk of Bleeding.
Brief Title: Safety and Effectiveness of Apixaban Compared to Warfarin in Patients With Non-valvular Atrial Fibrillation (a Type of Irregular Heart Rhythm) at Higher Chance of Bleeding
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661178
Record Dates: First submitted 2022-06-28; First posted 2022-07-22 (Actual); Results first posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Non-valvular Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

SUMMARY:
* The purpose of this study is to compare effectiveness and safety of warfarin and apixaban among non-valvular atrial fibrillation (NVAF) patients at higher chance of bleeding using a Japanese nation-wide administrative claims database.
* Atrial fibrillation (AF) is characterized by a fast, irregular heartbeat which can cause blood to pool in the atria and increase the chance of the formation of blood clots.
* An anticoagulation therapy is a critical treatment to prevent thromboembolism in NVAF patients.
* Apixaban was demonstrated superiority compared to warfarin in preventing stroke or systemic embolism, caused less bleeding, and resulted in lower mortality in patients with AF in Phase 3 clinical trial.
* Previously we have shown that bleeding risks as well as stroke/SE risks are less in real world clinical practice in Japan compared to warfarin. However there are limited apixaban data for Japanese NVAF patients with high bleeding risk(s).
* This study will evaluate the risk of stroke/systemic embolism as well as the risk of bleeding in the real world settings in Japanese patients with NVAF who has higher chance of bleeding

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with atrial fibrillation (AF) anytime in the baseline period or on the index date, also have definitive diagnosis of AF anytime in the baseline period, on the index date, or post-index period.
* Prescribed apixaban or warfarin on or after the day of AF diagnosis. The first observed prescription will be used to identify the patient's index date and treatment cohort
* No use of the any oral anticoagulants (OACs) during the baseline period (the 180 days before the index date)
* Age of 18 years or older on the index date

Exclusion Criteria:

* Having a diagnosis of valvular atrial fibrillation, post-operative atrial fibrillation, rheumatic atrial fibrillation or mechanical-valvular atrial fibrillation during the baseline and post-index period
* Having a procedure of prosthetic heart valve during the baseline period
* Having a cardiac surgery procedure record during the baseline period
* Having a diagnosis of venous thromboembolism during the baseline period
* Having a hemodialysis during the baseline period
* Female patients with pregnancy during the baseline and follow-up period
* Patients prescribed apixaban other than approved daily dose (<5 mg or >10 mg)
* Patients prescribed OACs during baseline period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study uses data from the MDV database, which includes the data used for both inpatient and outpatient insurance claims by hospitals according to the Diagnosis Procedure Combination (DPC) procedure.
  The study population will consist of adults with NVAF who are newly prescribed apixaban or warfarin.
Sampling Method: Probability Sample
Enrollment: 120722 (Actual)
Dates: Start 2022-08-25 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with non-valvular atrial fibrillation (NVAF) who were newly prescribed apixaban or warfarin with at least one high bleeding risk factor were observed in this retrospective observational study.
Pre-assignment Details: Data of eligible participants were extracted from Medical Data Vision Company Limited (MDV Co. Ltd.) database for duration of 01-Mar-2011 to 30-Jun-2021. Extracted data was evaluated for objectives of this study in approximately 1 month of this study.
Groups:
- Apixaban: Participants diagnosed with NVAF, who newly initiated apixaban, were included in this cohort. Data from 01-Mar-2011 to 30-Jun-2021, available in MDV database was observed retrospectively.
- Warfarin: Participants diagnosed with NVAF, who newly initiated warfarin, were included in this cohort. Data from 01-Mar-2011 to 30-Jun-2021, available in MDV database was observed retrospectively.
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 72095 | 48627
Completed | 72095 | 48627
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants whose data were extracted from database and observed in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 72095 | 48627 | 120722
Age, Customized [Count of Participants; unit: Participants]
  <= 64 years | 4471 | 4030 | 8501
  65-69 years | 4978 | 3855 | 8833
  70-79 years | 20621 | 14749 | 35370
  80-89 years | 33567 | 20677 | 54244
  =>90 years | 8458 | 5316 | 13774
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31786 | 19856 | 51642
  Male | 40309 | 28771 | 69080
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Composite Stroke and Systemic Embolism (SE) Events After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of composite stroke and SE events after index date was reported. Stroke events included the composite of any ischemic and any hemorrhagic stroke events (excluding non-traumatic extradural hemorrhage). Stroke after index date not including the index date was identified using hospital claims which had a stroke diagnosis code as the first listed International Classification of Diseases 10th Revision (ICD-10) diagnosis code. SE after index date not including the index date was identified using hospital claims which had a SE diagnosis code as the first listed ICD-10 diagnosis code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: Follow-up period during data observation period from Mar 2011 to Jun 2021 (approximately 10 years 4 months); extracted data evaluated in approximately 1 month of this study
Population: Eligible participants registered on MDV database, whose data was observed in the study. Analysis performed using Inverse probability treatment weighting (IPTW) method to balance participant characteristics among reporting groups. Here, "Overall Number of Participants Analyzed" is the number of participants after application of IPTW method to raw numbers and is different from the actual participants included in the reporting arm.
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Groups:
- Apixaban: Balanced Cohort: Participants diagnosed with NVAF, who newly initiated apixaban, were included in this cohort. Data from 01-Mar-2011 to 30-Jun-2021, available in MDV database was observed retrospectively. IPTW method was applied to balance the participants' characteristics.
- Warfarin: Balanced Cohort: Participants diagnosed with NVAF, who newly initiated warfarin, were included in this cohort. Data from 01-Mar-2011 to 30-Jun-2021, available in MDV database was observed retrospectively. IPTW method was applied to balance the participants' characteristics.
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 61.352 [59.413 to 63.354] | 75.078 [72.748 to 77.483]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p < 0.001, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.752, 95% CI 2-sided [0.719 to 0.787]

2. Primary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Major Bleeding Event After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of major bleeding event after index date was reported. Major bleeding was defined as any bleeding that required hospitalization for treatment. Major bleeding after index date was identified using hospital claims which had a bleeding diagnosis code as the first listed ICD-10 or disease code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: as for outcome 1
Population: Eligible participants registered on MDV database, whose data was observed in the study. Analysis performed using IPTW method to balance participant characteristics among reporting groups. Here, "Overall Number of Participants Analyzed" is the number of participants after application of IPTW method to raw numbers and is different from the actual participants included in the reporting arm.
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 16.788 [15.808 to 17.829] | 21.329 [20.138 to 22.590]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p < 0.001, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.747, 95% CI 2-sided [0.687 to 0.813]

3. Secondary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Ischemic Stroke Event After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of ischemic stroke event after index date was reported. Ischemic stroke after index date not including the index date was identified using hospital claims which had an ischemic stroke diagnosis code as the first listed ICD-10 diagnosis code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 49.038 [47.317 to 50.823] | 48.917 [47.071 to 50.835]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p < 0.001, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.909, 95% CI 2-sided [0.862 to 0.958]

4. Secondary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Hemorrhagic Stroke Event After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of hemorrhagic stroke event after index date was reported. Hemorrhagic stroke after index date not including the index date was identified using hospital claims which had a hemorrhagic stroke diagnosis code as the first listed ICD-10 diagnosis code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 9.384 [8.661 to 10.168] | 9.266 [8.498 to 10.104]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p = 0.378, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.948, 95% CI 2-sided [0.842 to 1.067]

5. Secondary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Systemic Embolism (SE) Event After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of SE event after index date was reported. SE after index date not including the index date was identified using hospital claims which had a SE diagnosis code as the first listed ICD-10 diagnosis code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 5.285 [4.750 to 5.882] | 18.923 [17.799 to 20.118]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p < 0.001, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.259, 95% CI 2-sided [0.229 to 0.294]

6. Secondary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Major Intracranial Bleeding Event After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of major intracranial bleeding event after index date was reported. Major intracranial bleeding after index date was identified using hospital claims which had an intracranial bleeding diagnosis code as the first listed ICD-10 or disease code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 14.490 [13.583 to 15.457] | 17.507 [16.436 to 18.649]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p < 0.001, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.767, 95% CI 2-sided [0.700 to 0.840]

7. Secondary Outcome: Incidence Rate Per 1000 Participant-Years For First Occurrence of Major Gastrointestinal (GI) Bleeding Event After Index Date: Balanced Cohorts
Description: Incidence rate per 1000 participant-years for the first occurrence of major GI bleeding event after index date was reported. Any GI bleeding after index date was identified using hospital claims which had a GI bleeding diagnosis code as the first listed ICD-10 or disease code. Index date: date when participants initiated warfarin or apixaban. Follow-up period: from next day of the index date till occurrence of target outcome event, discontinuation of apixaban or warfarin; switching from apixaban or warfarin; withdrawal from the database, whichever occurred first.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 1000 Participant-Years
Arm/Group | Apixaban: Balanced Cohort | Warfarin: Balanced Cohort
Number analyzed (Participants) | 72141 | 48619
Events Per 1000 Participant-Years | 36.836 [35.354 to 38.380] | 36.943 [35.350 to 38.607]
Statistical Analysis 1: Comparison: Apixaban: Balanced Cohort vs Warfarin: Balanced Cohort; Test type: Other; p = 0.022, COX Proportional Hazards Regression; Hazard Ratio (HR) = 0.932, 95% CI 2-sided [0.877 to 0.990]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected during the study
Description: This study involved data that existed as structured data by the time of study start. In these data sources, individual participants data was not retrieved or validated, and it was not possible to link (i.e., identify a potential association between) a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) (i.e., identifiable patient, identifiable reporter, a suspect product, and event) could not be met.
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/05/NCT05471505/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/05/NCT05471505/SAP_001.pdf